CLINICAL TRIAL: NCT00978172
Title: A Phase IV Study on the Safety and Effectiveness of a Fixed-dose Combination of Artesunate and Mefloquine (Artequin[TM] Paediatric) Administered for 3 Days in Children With Uncomplicated Plasmodium Falciparum Malaria in Africa
Brief Title: Safety and Efficacy Study of Artesunate and Mefloquin in Children With Uncomplicated Malaria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mepha Ltd. (Industry)
Collaborators: Centre Mère et Enfant de la Fondation Chantal Biya (Other)
Responsible Party: Prof. Dr. Félix Tietche, Department of Paediatry, Medical faculty, University of Yaounde (Cameroun)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ART-P 001-2007
Record Dates: First submitted 2009-09-10; First posted 2009-09-16 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artesunate; Mefloquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: artesunate and mefloquine — artesunate (50 mg/day) and mefloquine (125 mg/day) fixed dose formulation (stick pack) once daily for 3 consecutive days, orally
  Other Names: Artequin[TM] Paediatric stickpack

SUMMARY:
The present study aims to investigate and to assess possible neurological and neuropsychiatric events in young children in west Africa with uncomplicated P. falciparum malaria after a 3-day treatment of Artequin Paediatric under "real life conditions."

DETAILED DESCRIPTION:
The study aims investigating the safety profile of Artequin Paediatric in a 3-day treatment of children with uncomplicated P. falciparum malaria under "real life conditions" in West Africa. Important parameters, such as concomitant medication, the patient's medical history and diseases, differential WBC counts, the presence of parasitaemia as well as the patient's compliance are evaluated. Detailed recording of possible AEs and SAEs enable additionally an assessment of the safety and effectiveness of Artequin Paediatric over a period of 63 days following treatment initiation. The present study primarily serves to detect and assess possible neuropsychiatric and neurological events in young children using a standardized questionnaire and axamination.

ELIGIBILITY:
Inclusion Criteria:

* Body weight from ≥ 10 kg to ≤ 20 kg.
* Presence of acute uncomplicated P. falciparum malaria with a diagnosis confirmed by a positive blood smear with asexual forms of P. falciparum only.
* Counts of asexual forms of P. falciparum: 2'000 to 250'000 parasites per µL of blood.
* Presence of fever defined as axillary temperature of ≥37.5 °C (≥ 38 °C if oral, rectal or tympanic temperature) or a history of fever within the last 24 hours.
* Written informed consent provided by the patient and parent or guardian. If the person is unable to write, thumb print witnessed consent is permitted.
* Willingness and ability of the patient and the parent or guardian to comply with study protocol for the duration of the study.
* Patients who are able to take oral medication.

Exclusion Criteria:

* Patients with severe/complicated malaria as defined by the World Health Organization, 2000, Severe falciparum malaria (18).
* Known history or evidence of clinically significant disorders: neurological, psychiatric (depression, psychosis or schizophrenia), cardiovascular (including arrhythmia), pulmonary, metabolic, gastrointestinal, endocrine diseases or malignancies.
* Patients with a history of epilepsy or of convulsions.
* Patients who received any anti-malarial treatment within 7 days prior to enrolment including any substance with anti-malarial activity, e.g. antibiotics)or treatment with mefloquine within 30 days prior to enrolment.
* Patients with a hypersensitivity or allergic reaction to artemisinins or mefloquine or any chemically related entity (e.g. quinine).
* Patients who participated in any investigational drug trial within 30 days prior to enrolment.
* Patients with vomiting 3 or more times within 24 hours of enrolment or more than 3 copious liquid stools within 24 hours.
* Patients with known renal impairment.
* Patients who do require parenteral treatment.
* Patients who have had a splenectomy.
* Known immunocompromised patients and who are receiving immunosuppressive agents and/or patients with known human immunodeficiency virus (HIV) infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2007-12; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the neuropsychiatric and neurological safety of a fixed-dose combination of artesunate and mefloquine (Artequin Paediatric) in the treatment of children (>=10kg to <=20kg body weight) with uncomplicated P. falciparum malaria | Baseline (day1), day 7, day 28, day 63

SECONDARY OUTCOMES:
To determine further safety and effectiveness parameters of Artequin Paediatric | Baseline (day1), day 4, day7, day 28, day 63

CONTACTS AND LOCATIONS:
Overall Officials: Felix Tietche, Prof, Principal Investigator — Faculty of Medicine and Biomedical Sciences University of Yaounde (Cameroon)
Locations (1):
- Centre Mère et Enfant, Fondation Chantal Biya, Yaoundé, Yaounde, Cameroon